CLINICAL TRIAL: NCT06852157
Title: Evaluation Of The Diagnostic And Prognostic Value Of Immunohistochemical Markers In Precancerous Lesions Of The Cervix
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cervix-IHC
Record Dates: First submitted 2024-12-01; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cervix Cancer
Keywords: cervix cancer; gynaecology
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Histocompatibility Testing; Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with precancerous lesions of the cervix CIN/SIL (Other): Patients diagnosed with precancerous lesions of the cervix CIN/SIL undergoing diagnostic biopsy/uterine conization since January 2000
  Interventions: Diagnostic Test: Tissue, diagnostic and prognostic accuracy

INTERVENTIONS:
Diagnostic Test: Tissue, diagnostic and prognostic accuracy — The clinical data and histological samples of patients with a diagnosis of CIN/SIL on cervical biopsies or conization (performed as required by the normal procedure) will be consecutively acquired from all those taken at the Operative Unit of Gynaecology and Physiopathology of Human Reproduction starting from January 2000 and stored at the Operative Unit of Pathological Anatomy and Histology.
  Samples fixed in neutral buffered formalin and paraffin added at 50°C will be analysed by repeating histological examination and performing immunohistochemistry for BAG3. All analyses will be performed blinded to the clinical data of the patients and the results of the original examinations. No patients will be examined ex novo, as only paraffin-embedded tissue samples obtained at the time of the initial diagnosis will be analysed.

SUMMARY:
The study aims to evaluate the expression of certain proteins and their diagnostic and prognostic value in precancerous lesions of the cervix.

DETAILED DESCRIPTION:
Cervical cancer is the second most common malignancy in women and the most common gynaecological cancer worldwide. Numerous risk factors are associated with the development of cervical cancer; in particular, human papilloma virus (HPV) infection plays a decisive role in the development of the neoplasm. Almost all cervical cancers are caused by persistent human papilloma virus (HPV) infections.

In particular, squamous cell carcinoma accounts for about 70% of cervical cancers; its precursor is called 'cervical intraepithelial neoplasia' (CIN) or 'squamous intraepithelial lesion' (SIL) and is classified according to the degree of dysplasia. The 'CIN' classification system defines three categories: CIN1 (dysplasia limited to the lower third of the epithelium), CIN2 (dysplasia extending into the middle third of the epithelium) and CIN3 (dysplasia extending into the upper third of the epithelium). More recently, the 'CIN' system has been replaced by the 'SIL' system, which appears more reproducible and biologically relevant. The 'SIL' system reduces the categories from three to two: low grade - SIL (L - SIL, overlapping CIN1) and high grade - SIL (H - SIL, grouping CIN2 and CIN3 together).

Several diagnostic markers have been proposed, such as athanogene 3 associated with Bcl - 2 (BAG3) and others with prognostic value such as topoisomerase 2A (TOP2), minichromosome maintenance protein 2 (MCM 2), Ki-67, P16INK4, P-53 associated with cervical cancer. However, there is no strong evidence for the association of these markers with precancerous lesions.

Our study therefore aims to investigate the diagnostic and prognostic value of Bcl-associated athanogene 3 - 2 (BAG3) in patients diagnosed with CIN/SIL undergoing colposcopic cervical biopsies or conization.

This clinical trial is therefore a tissue-based, diagnostic and prognostic accuracy, retrospective cohort, single-center, non-profit, pilot study and foresees that histological sections obtained at the time of initial diagnosis will be re-evaluated in blinded fashion by two pathologists regarding histological diagnosis, histotype, histological grading, lymphocytic infiltrate. They will then be subjected to immunohistochemistry according to the specific protocol for BAG3.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of CIN/SIL undergoing cervical biopsy/concussion whose tissue sample is archived at the Operative Unit of Pathological Anatomy and Histology
* Obtaining written informed consent for the use of biological samples
* Patients aged 18 years and over

Exclusion Criteria: none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Expression of BAG3 | enrollment through study completion, an average of 1 year
  Expression of BAG3 in patients diagnosed with precancerous lesions of the cervix

SECONDARY OUTCOMES:
Correlation between BAG3 expression and the degree of dysplasia of cervical lesions | After enrollment, through study completion, an average of 1 year
  Correlation between BAG3 expression and the degree of dysplasia of cervical lesions
Evolution of bag3 expression over time | After enrollment, through study completion, an average of 1 year
  Evolution of BAG3 expression over time in patients with cervical biopsies/concussions afterwards

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Casadio, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy